CLINICAL TRIAL: NCT05715294
Title: TC Gazi University
Brief Title: The Effect of Music on Sleep Quality in Behçet's Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Özlem Canbolat, Assistant Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ozlem Canbolat
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Sleep Quality; Behçet Disease
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Behcet Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Application Group (Experimental): After explaining the purpose of the study and the way it was applied to behçet's patients in the music group, Introductory Information Form, Behçet's Syndrome Activity Scale (BSAS), Richards-Campbell Sleep Questionnaire (RCSQ) will be applied. Patients will listen to music composed in Uşşak makam for 50 minutes before going to bed every day for 7 days. After the first interview, the patients will be reminded of the music application by phone call and 2 text messages every day by the researcher. Interviews will be recorded on the Patient's Telephone Follow-up Form while Listening to Music. On the 8th day, the BSAS and RCSQ scales will be reapplied to the patients in the intervention group.
  Interventions: Other: Music Application
- Control Group (No Intervention): After explaining the purpose of the study and the way it was applied to behçet's patients in the control group, Introductory Information Form, Behçet's Syndrome Activity Scale (BSAS), Richards-Campbell Sleep Questionnaire (RCSQ) will be applied.No application will be made to the control group. On the 8th day, the BSAS and RCSQ scales will be reapplied to the patients.

INTERVENTIONS:
Other: Music Application — A music CD was prepared within the scope of passive music listening practice. To determine the music, the researcher advice and literature knowledge of Turkish Music A music CD was prepared within the scope of passive music listening practice. To determine the music, the researcher advice and literature knowledge of Turkish Music Research and Promotion Society (TUMATA) was used. In the music application, the selecting instrumental music (ussak maqam which is Turkish Music Maqam) was used. The prepared Music CD will be played on the phones of patients with android processor phones. Patients will be told that they should listen to the music lying down and in a comfortable position, and that they should not use headphones while listening to music. Before going to bed, the patients will be listened to music composed in Ussak maqam for 50 minutes every day for 7 days.
  Arms: Music Application Group

SUMMARY:
The aim of this study was to evaluate effect of music on sleep quality in patients with Behçet's disease. The population of the study consists of behçet patients who applied to the Rheumatology outpatient clinic of Medical Faculty Hospital, who met the research criteria and agreed to participate in the study.

The study will conduct in a randomized controlled experimental design with two groups. The sample of the study will be 50 behçet patients the music practice group (25) and the control group (25). The research will be carried out between December 2022 and December 2023. In this study, data will with collect Descriptive Information Form, Behçet's Syndrome Activity Scale (BSAS) and Richard-Campbell Sleep Scale (RCUI).

DETAILED DESCRIPTION:
This study will be conducted as a parallel group randomized controlled experimental study to determine the effect of listening to music in the uşşak makam on sleep quality in Behçet's Diseases.The population of the research will be Behçet's patients receiving outpatient treatment in the Rheumatology outpatient clinic of a university hospital.G.Power program was used to calculate the sample size of the study. In descriptive studies, the t tests - Means: Difference between two independent means (two groups) model was used to determine the sample size when the number of individuals in the universe was not known. While determining the sample volume in the research, the test for the main hypothesis was determined at the first stage and the required averages were obtained from Bakır's research in 2019, which is compatible with our study in the literature (Bakır, 2019). According to the g-power analysis, with 95% confidence level and α=0.05 margin of error, it has an effect size of 0.941 and a tolerance ratio of 5%; In this study, the power of the test was determined as p: 0.05, (1-β): 90%, t = 2.015, and in line with this information, it was concluded that the number of samples required for the study was 46 people in both groups. Considering the possible losses from the experimental study, the number of samples was increased by 10% and it was decided that the total sample size would be 50 people, 25 people in the intervention group and 25 people in the control group.Application In this study, intervention and control groups will be studied in a pre-test and post-test design. No intervention will be applied to the control group. Passive music listening practice for the intervention group.

ELIGIBILITY:
Inclusion Criteria:

18 years or older Having been diagnosed with Behçet's Disease for at least 6 months A score of 0-25 on the Richard-Campbell Sleep Questionnaire No visual or hearing impairment Being literate Ability to understand and speak Turkish Having mental and cognitive competence Not having a psychiatric diagnosis It is voluntary to participate in the study. Not using sleeping pills Become an Android processor phone

-

Exclusion Criteria:

Unreachable during phone calls with sleep apnea Chronic diseases that can affect sleep such as COPD, Asthma, Heart failure not continuing research Patients using sleeping pills

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Richard - Campbell Sleep Questionnaire | a day before the music application
  Scores from the scale range from 0 to 100, and the higher the score, the higher the sleep quality. "0-25" points poor sleep quality, "76-100" points good sleep quality.
Richard - Campbell Sleep Questionnaire | after music application, 8th day
  Scores from the scale range from 0 to 100, and the higher the score, the higher the sleep quality. "0-25" points poor sleep quality, "76-100" points good sleep quality.

IPD SHARING:
Plan to Share IPD: Undecided